CLINICAL TRIAL: NCT00199004
Title: German Multicenter Trial for Treatment Optimisation in Acute Lymphoblastic Leukemia in Adults and Adolescents Above 15 Years With Rituximab for Improvement of Prognosis in CD20 Positive Standard Risk ALL (Amend 2)
Brief Title: Trial for Treatment of Adult Patients With Standard Risk Acute Lymphoblastic Leukemia With Chemotherapy and Rituximab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMALL03
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2008-05

CONDITIONS: Adult Acute Lymphocytic Leukemia
Keywords: ALL; Treatment; De novo; Minimal residual disease; Rituximab; Adult
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — Cyclophosphamide; Dexamethasone; Prednisolone; Vincristine; Daunorubicin; Asparaginase; Methotrexate; Cytarabine; Mercaptopurine; Granulocyte Colony-Stimulating Factor; Vindesine; Etoposide; Doxorubicin; Thioguanine; Teniposide; Rituximab; Stem Cell Transplantation

INTERVENTIONS:
Drug: Cyclophosphamide
Drug: Dexamethasone / Prednisolone
Drug: Vincristine
Drug: Daunorubicin
Drug: Asparaginase
Drug: Methotrexate
Drug: Cytarabine
Drug: Mercaptopurine
Drug: G-CSF
Drug: Vindesine
Drug: VP16
Drug: Adriamycin
Drug: Thioguanine
Drug: VM26
Drug: Rituximab
Procedure: CNS irradiation
Procedure: Mediastinal irradiation (if residual TU)
Procedure: Stem cell transplantation

SUMMARY:
The study evaluates the efficacy and tolerability of an intensified induction and consolidation therapy in combination with rituximab in CD20 positive standard risk patients. Thereafter patients receive additional consolidation and reinduction cycles combined with rituximab. In parallel minimal residual disease is evaluated. After six months and one year the decision on intensification or discontinuation of therapy is made based on results of MRD evaluation

ELIGIBILITY:
Inclusion Criteria:

* B-precursor ALL (common / pre B-ALL)
* Standard risk
* CD20 expression >20%
* Ph/BCR-ABL negative
* Age 15-65 years (55-65 if biologically younger)
* Written informed consent

Exclusion Criteria:

* Severe complications due to leukemia or secondary illnesses
* Late relapse of childhood ALL
* Cytostatic pretreatment
* Pregnancy
* Severe psychiatric illness or other circumstances which may compromise cooperation of the patient or informed consent
* Known severe allergy to foreign proteins

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Remission rate (cytologic, Remission rate (molecular), Remission duration, Disease free survival, Overall survival

SECONDARY OUTCOMES:
Dose and time compliance, Toxicity according to WHO, Death in induction and CR, Course of MRD

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hoelzer, MD,PhD, Study Chair — University Hospital, Medical Dept. II
Locations (1):
- University Hospital of Frankfurt, Medical Dept. II, Frankfurt, Germany

REFERENCES:
- See also: German Leukemia Trial Registry — http://www.studienregister-online.de